CLINICAL TRIAL: NCT06915753
Title: A Multicenter, Open-label, First-in-Human Study of TYRA-430 in Advanced Hepatocellular Carcinoma and Other Solid Tumors With Activating FGF/FGFR Pathway Aberrations
Brief Title: Safety and Preliminary Anti-Tumor Activity of TYRA-430 in Advanced Hepatocellular Carcinoma and Other Solid Tumors With Activating FGF/FGFR Pathway Aberrations
Acronym: SURF431
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYR430-101
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Hepatocellular Carcinoma; Solid Tumors; Solid Tumor, Adult; FGFR Gene Amplification; FGFR Gene Alterations; FGFR3 Gene Alteration; FGFR3 Gene Mutation; Advanced Solid Tumors; FGFR4 Gene Mutation; FGFR4 Gene Fusions; FGF19 Gene Amplification; FGF19 Gene Overexpression; FGFR3 Gene Fusions; Locally Advanced Unresectable Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; metastatic cancer; solid tumors; FGF19 gene amplifications; FGFR4 gene alterations; FGFR3 gene alterations; FGF19 gene alterations; FGFR4 gene mutations; FGFR4 gene fusions; FGFR3 gene mutations; FGFR3 gene fusions; FGF19 gene overexpression; locally advanced unresectable cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Dose Escalation (Experimental): Dose escalation of TYRA-430 as monotherapy at various dose levels.
  Interventions: Drug: TYRA-430
- Part B - Cohort 1 Dose Expansion (Experimental): Dose expansion group for TYRA-430 monotherapy in advanced HCC at a dose(s) determined in Part A.
  Interventions: Drug: TYRA-430
- Part B - Cohort 2 Dose Expansion (Experimental): Dose expansion group for TYRA-430 monotherapy in advanced solid tumors at a dose(s) determined in Part A.
  Interventions: Drug: TYRA-430

INTERVENTIONS:
Drug: TYRA-430 — Oral TYRA-430 given daily.

SUMMARY:
A Phase 1 study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamic (PD), and preliminary antitumor activity of TYRA-430 in cancers with FGF/FGFR pathway aberrations, including locally advanced/metastatic hepatocellular carcinoma and other advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, first-in-human, Phase 1 global study of TYRA-430, a first-in-class, selective, reversible fibroblast growth factor receptor (FGFR) 4 and 3 inhibitor, in locally advanced/metastatic hepatocellular carcinoma and other advanced solid tumors that contain FGF/FGFR pathway aberrations.

ELIGIBILITY:
Key Inclusion Criteria:

All Patients:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* Adequate end organ function.
* Ability to swallow oral formulations.
* Ability to understand and willingness to sign the ICF.

Part A:

* Histologically confirmed locally advanced unresectable/metastatic HCC or histologically confirmed advanced solid tumor with documented FGF/FGFR pathway alterations
* For participants with histologically confirmed locally advanced or metastatic HCC:

  * Barcelona Clinic Liver Cancer (BCLC) stage B that is not eligible for locoregional therapy, or stage C.
  * Child-Pugh Score class A
* Must have previously received SOC appropriate for their tumor type. Any number of prior therapies, including FGFR inhibitors, are permitted.
* Agree to provide archival tumor tissue no older than 2 years from the time of enrollment, if available. If an archived specimen is not available, a biopsy is not required.

Part B, Cohort 1:

* Histologically confirmed locally advanced/metastatic HCC who have previously received standard of care.
* Barcelona Clinic Liver Cancer (BCLC) stage B that is not eligible for locoregional therapy, or stage C.
* Child-Pugh Score class A
* Availability of an archival formalin-fixed paraffin-embedded (FFPE) tumor tissue specimen obtained ≤2 years prior to screening for submission to sponsor-designated central laboratory for FGF19 IHC testing.
* At least 1 measurable lesion by RECIST v1.1.

Part B, Cohort 2:

* Histologically confirmed advanced solid tumor except FGFR3-altered urothelial carcinoma and primary central nervous system tumors who have previously received standard of care. Note: Participants with confirmed diagnosis of locally advanced or metastatic HCC are not eligible for Cohort 2.
* Must have an eligible activating gain-of-function alteration in the FGFR3 or FGFR4 gene, or focal amplifications of FGF19
* Archival tumor tissue biopsy specimen no older than 2 years from the time of enrollment, if available. If a tissue biopsy specimen is not available, a biopsy is not required.
* At least 1 measurable lesion by RECIST v1.1.

Key Exclusion Criteria:

All Patients:

* Have disease that is suitable for local therapy administered with curative intent.
* Have not recovered from reversible toxicity of prior anticancer therapy to < Grade 1 or baseline (except toxicities that are not clinically significant or not expected to resolve, including but not limited to, alopecia, fatigue, skin discoloration, or Grade 1 neuropathy).
* Have received the following anticancer therapy:

  1. Any immunotherapy or other antibody therapy within 28 days prior to the first dose of the study drug.
  2. A TKI < 5 days or 5X the terminal Phase elimination half-lives, whichever is longer, prior to the first dose of TYRA-430.
  3. Other systemic therapy not listed above < 14 days prior to the first dose of the study drug.
* Participant discontinued a prior anti-FGFR therapy due to significant toxicity, defined as hepatotoxicity ≥ Grade 3 or any Grade 4 toxicity according to CTCAE v5.0.
* Has a serum phosphorus level > upper limit of normal (ULN) during screening that remains >ULN despite medical management.
* History of or current uncontrolled cardiovascular disease.
* Active, symptomatic, or untreated brain metastases.
* Have a diagnosis of primary CNS malignancies.
* Gastrointestinal disorders that will affect oral administration or absorption of TYRA-430.
* Females who are pregnant, breastfeeding, or planning to become pregnant and males who plan to father a child while enrolled in this study.
* Any reason that, in the view of investigator, would substantially impair the ability of the participant to comply with study procedures and increase the risk to the participant.

Part B, Cohort 1:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Prior treatment with pan-FGFR inhibitors or FGFR4-selective inhibitors.

Part B, Cohort 2:

* Histologically confirmed locally advanced/metastatic HCC.
* Histologically confirmed urothelial cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 1 year
  MTD determination: dose limiting toxicity (DLT) rate in the first 28-day cycle
Rate and severity of adverse events of TYRA-430 as monotherapy | First dose of study drug through 28 days after the last dose of study drug
  Number of participants with TEAEs as assessed by CTCAE, v5.0
Recommended Phase 2 dose(s) of TYRA-430 | Up to 2 years
  To determine recommended Phase 2 dose(s) of TYRA-430

SECONDARY OUTCOMES:
Cmax | Up to 2 years
Tmax | Up to 2 years
AUC0-last | Up to 2 years
AUCTau | Up to 2 years
AUC0-∞ | Up to 2 years
Vd/F | Up to 2 years
CL/F | Up to 2 years
t1/2 | Up to 2 years
Overall Response Rate (ORR) | Up to 3.5 years
  The proportion of patients who experience a best response of confirmed CR or PR per RECIST 1.1
Duration of Response (DOR) | Up to 3.5 years
  Time from first investigator-assessed response to radiographic disease progression or death.
Disease Control Rate (DCR) | Up to 3.5 years
  Best response of CR, PR, or SD per RECIST v1.1 > 12 months.
Time to Response (TTR) | Up to 3.5 years
  The median time from the start of therapy to first response in confirmed responders.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, MD, Study Chair — Tyra Biosciences, Inc
Locations (16):
- United States (9):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center at Mount Zion, San Francisco, California
  - Stanford Cancer Institute, Stanford, California
  - The University of Kansas Medical Center, Westwood, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Mass General Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University Irving Medical Center, New York, New York
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
- University Health Network Princess Margaret Cancer Center, Toronto, Ontario, Canada
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided